CLINICAL TRIAL: NCT00660673
Title: Open-Label Continuation Treatment Study With Levodopa - Carbidopa Intestinal Gel In Subjects With Advanced Parkinson's Disease And Severe Motor-Fluctuations Who Have Exhibited A Persistent And Positive Effect To Treatment In Previous Studies
Brief Title: Open Label Continuation Treatment Study With Levodopa-Carbidopa Intestinal Gel in Advanced Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: IQVIA, formerly Quintiles (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S187.3.005; 2008-001329-33 (EudraCT Number)
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Advanced Parkinson's Disease
Keywords: levodopa/carbidopa intestinal gel; Severe Motor Fluctuations; Levodopa; Carbidopa; Parkinson's Disease; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levodopa-Carbidopa Intestinal Gel (Experimental): Initial dosing is based on the dosing regimen that the participant received during the previous LCIG study. Dosing is individually optimized and can be adjusted at any time during the study as clinically indicated. The total dose/day of LCIG is composed of 3 individually adjusted doses. The morning dose is administered as a bolus infusion, usually 5 to 10 mL (100 to 200 mg levodopa). The maintenance dose is adjustable in steps of 2 mg/hour (0.1 mL/hour), within a range of 1 to 10 mL/hour (20 to 200 mg levodopa/hour) and is usually 2 to 6 mL/hour (40 to 120 mg levodopa/hour). Participants will be allowed to self-administer extra doses of LCIG to address immediate medical needs, normally 0.5 to 2.0 mL.
  Participants will receive LCIG until it is commercially available.
  Interventions: Drug: Levodopa-Carbidopa Intestinal Gel (LCIG); Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: Percutaneous Endoscopic Gastrostomy with jejunal extension tube (PEG-J)

INTERVENTIONS:
Drug: Levodopa-Carbidopa Intestinal Gel (LCIG) — LCIG for upper-intestinal infusion is a suspension of levodopa (20 mg/mL) and carbidopa (5 mg/mL) in an aqueous gel that is dispensed in a medication cassette reservoir containing 100 mL of LCIG.
  Other Names: Carbidopa-Levodopa Enteral Suspension (CLES); Duopa®; Duodopa®
Device: CADD-Legacy® 1400 ambulatory infusion pump — Portable infusion pump (CADD-Legacy Pump Model 1400) connected to the LCIG medication cassette reservoir.
Device: Percutaneous Endoscopic Gastrostomy with jejunal extension tube (PEG-J) — All participants previously had a PEG-J placed in one of the prior LCIG studies.

SUMMARY:
The primary objective of this study is to provide continued access to levodopa-carbidopa intestinal gel (LCIG), to participants who have already participated in an open-label efficacy and safety study with the same treatment (Study S187.3.003 [NCT00360568] or Study S187.3.004 [NCT00335153]).

ELIGIBILITY:
Inclusion Criteria:

* The participant should have completed participation in Study S187.3.003 or S187.3.004; and, in the opinion of the Principal Investigator, would benefit from long-term treatment with LCIG.
* For Canada, participants will be allowed to participate in the S187.3.005 study with a minimum of 6 months of exposure to LCIG in the S187.3.004 study.
* The participant must be able to understand the nature of the study and must provide written informed consent prior to the conduct of any study related procedures. If the participant does not have the capacity to provide informed consent, full informed consent must be obtained from the participant's legally authorized representative. Consenting will be performed according to local regulations.

Exclusion Criteria:

* Medical, laboratory, psychiatric, or surgical issues deemed by the investigator to be clinically significant and which could interfere with the participant's participation in the study.

Ages: 30 Years to 99 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2009-11-13 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (61):
- United States (31):
  - University of Alabama at Birmingham /ID# 49941, Birmingham, Alabama
  - The Research Center of Southern California /ID# 49928, Encinitas, California
  - The Parkinson's & Movement Disorder Institute - Fountain Valley /ID# 49915, Fountain Valley, California
  - Universtiy of Southern California /ID# 49913, Los Angeles, California
  - Colorado Neurological Institute /ID# 49927, Englewood, Colorado
  - Georgetown University Hospital /ID# 49931, Washington D.C., District of Columbia
  - Bradenton Research Center, Inc /ID# 49929, Bradenton, Florida
  - Neurologic Consultants, PA /ID# 49918, Fort Lauderdale, Florida
  - University of Florida - Archer /ID# 49935, Gainesville, Florida
  - University of Florida /ID# 49922, Jacksonville, Florida
  - Charlotte Neurological Service /ID# 49916, Port Charlotte, Florida
  - University of South Florida /ID# 49919, Tampa, Florida
  - Georgia Regents University /ID# 49938, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 49944, Chicago, Illinois
  - Rush University Medical Center /ID# 49930, Chicago, Illinois
  - University of Kentucky Chandler Medical Center /ID# 49940, Lexington, Kentucky
  - Louisiana State Univ HSC /ID# 49945, Shreveport, Louisiana
  - Univ Maryland School Medicine /ID# 49934, Baltimore, Maryland
  - Johns Hopkins University /ID# 49937, Baltimore, Maryland
  - Washington University-School of Medicine /ID# 49933, St Louis, Missouri
  - University of Nebraska Medical Center /ID# 49911, Omaha, Nebraska
  - North Shore University Hospital /ID# 49932, Manhasset, New York
  - The Mount Sinai Hospital /ID# 49942, New York, New York
  - Columbia Univ Medical Center /ID# 49943, New York, New York
  - Raleigh Neurology Associates /ID# 49923, Raleigh, North Carolina
  - Wake Forest Univ HS /ID# 49939, Winston-Salem, North Carolina
  - University of Cincinnati /ID# 49914, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 76173, Cleveland, Ohio
  - University of Vermont Medical Center /ID# 49912, Burlington, Vermont
  - King County Public Hospital /ID# 49917, Kirkland, Washington
  - Froedtert Memorial Lutheran Hospital /ID# 49924, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital /ID# 50081, Westmead, New South Wales
  - Royal Adelaide Hospital /ID# 50083, Adelaide, South Australia
  - Austin Hospital /ID# 50082, Heidelberg, Victoria
- Canada (3):
  - University of Alberta /ID# 78476, Edmonton, Alberta
  - Toronto Western Hospital /ID# 75913, Toronto, Ontario
  - CHUM - Notre-Dame Hospital /ID# 74513, Montreal, Quebec
- Czechia (5):
  - Fakultni Nemocnice u Svate Anny /ID# 50085, Brno
  - Fakultni nemocnice Hradec Kralove /ID# 50088, Hradec Králové
  - Pardubicka krajska nemocnice, a.s., Pardubice
  - Vseobecna fakultni nemocnice v Praze /ID# 50086, Prague
  - Fakultni Nemocnice v Motole /ID# 50084, Prague
- Tel Aviv Sourasky Medical Center /ID# 50089, Tel Aviv, Israel
- New Zealand (4):
  - Waikato Hospital /ID# 50091, Hamilton, Waikato Region
  - Auckland City Hospital /ID# 50093, Auckland
  - New Zealand Brain Research Institute/ID# 50090, Christchurch
  - Wellington Hospital /ID# 50092, Wellington
- Poland (2):
  - NZOZ Centrum Medyczne HCP /ID# 50094, Poznan, Greater Poland Voivodeship
  - Miejskie Centrum Medyczne im. dr. Karola Jonschera w Lodzi /ID# 50096, Lodz, Łódź Voivodeship
- Portugal (3):
  - Hospitais da Universidade de Coimbra /ID# 50098, Coimbra
  - Hospital de Santa Maria /ID# 50099, Lisbon
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 50101, Porto
- Russia (5):
  - Scientific Research Medical Complex Your Health /ID# 50104, Kazan'
  - Institution of the Russian Academy of Medical Sciences Scientific Centre of Neurology /ID# 50102, Moscow
  - Military Medical Academy n.a. Kirov /ID# 50103, Saint Petersburg
  - I.P. Pavlov First St. Petersburg State Medical University /ID# 50107, Saint Petersburg
  - City Clinical Hospital #40 /ID# 50106, Saint Petersburg
- Thailand (2):
  - King Chulalongkorn Mem Hosp /ID# 50108, Bangkok
  - Siriraj Hospital /ID# 50109, Bangkok
- United Kingdom (2):
  - The Walton Centre NHS Foundation /ID# 50003, Liverpool
  - National Hospital for Neurology & Neurosurgery, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Result] Fernandez HH, Boyd JT, Fung VSC, Lew MF, Rodriguez RL, Slevin JT, Standaert DG, Zadikoff C, Vanagunas AD, Chatamra K, Eaton S, Facheris MF, Hall C, Robieson WZ, Benesh J, Espay AJ. Long-term safety and efficacy of levodopa-carbidopa intestinal gel in advanced Parkinson's disease. Mov Disord. 2018 Jul;33(6):928-936. doi: 10.1002/mds.27338. Epub 2018 Mar 23. PMID 29570853
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in November 2009 and was completed in October 2012. Participants were enrolled at 61 sites in 11 countries: Australia, Canada, Czech Republic, Israel, New Zealand, Poland, Portugal, the Russian Federation, Thailand, the United Kingdom, and the United States.
Pre-assignment Details: This study was an open-label extension study for participants with Parkinson's disease (PD) who had completed one of the prior studies S187.3.003 (NCT00360568) or S187.3.004 (NCT00335153). Participants were to receive continued access to levodopa-carbidopa intestinal gel (LCIG) in the extension study until treatment became commercially available in their home country.
Groups:
- Levodopa-Carbidopa Intestinal Gel: Participants received levodopa-carbidopa intestinal gel (LCIG), continuously administered through a percutaneous endoscopic gastrostomy with jejunal extension tube (PEG-J) directly into the jejunum via a portable pump during 16 hours of wakefulness.
  Initial dosing was based on the dosing regimen that the participant received during the previous LCIG study. Dosing was individually optimized and adjusted as clinically indicated.
  In addition to a morning dose (to prime the intestinal tube and rapidly achieve the therapeutic dose level) of 5 to 10 mL (100 to 200 mg levodopa), and the continuous infusion usually 2 to 6 mL/hour (40 to 120 mg levodopa/hour), participants were allowed to self-administer additional doses of LCIG to address immediate subjective needs (eg, deterioration of motor function).
  Participants received LCIG until it became commercially available.
Period: Overall Study
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Started | 262
Completed | 145
Not Completed | 117
Not completed — Adverse Event | 84
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 22
Not completed — Administrative | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Levodopa-Carbidopa Intestinal Gel: Participants received LCIG continuously administered through a PEG-J directly into the jejunum via a portable pump during 16 hours of wakefulness.
  Initial dosing was based on the dosing regimen that the participant received during the previous LCIG study. Dosing was individually optimized and adjusted as clinically indicated.
  In addition to a morning dose (to prime the intestinal tube and rapidly achieve the therapeutic dose level) of 5 to 10 mL (100 to 200 mg levodopa), and the continuous infusion usually 2 to 6 mL/hour (40 to 120 mg levodopa/hour), participants were allowed to self-administer additional doses of LCIG to address immediate subjective needs (eg, deterioration of motor function).
  Participants received LCIG until it became commercially available.
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.9)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 133
  ≥ 65 years | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 255
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 21
  Black of African Heritage or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 239

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) which started on or after the date of the first LCIG Infusion in this study and within 30 days of the date of the last PEG-J exposure.
  At least possibly drug-related is defined as TEAEs assessed as having a "Possible" or "Probable" or missing relationship to study drug.
  Serious AEs included any untoward medical occurrence that:
  * Resulted in death
  * Was life-threatening
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * was a congenital anomaly/birth defect
  The severity of all AEs was characterized as mild, moderate or severe according to the following definitions:
  * Mild: usually transient and do not interfere with daily activities.
  * Moderate: low level of inconvenience or concern to the subject, may interfere with daily activities.
  * Severe: events interrupt the subject's usual daily activity.
Time Frame: From first dose of LCIG in this study up to 30 days after the date of last PEG-J exposure; median duration of treatment was 1178 days, with a maximum of 4217 days (11.5 years).
Population: All participants who received LCIG in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Participants
  Any treatment-emergent adverse event (TEAE) | 253
  TEAE at least possibly related to study drug | 219
  Serious TEAE | 159
  Severe TEAE | 152
  TEAE leading to premature study discontinuaton | 82
  TEAE leading to death | 58

2. Secondary Outcome: Number of Participants With Device Complications
Description: Device complications include complications with the pump, intestinal tube, PEG-J or stoma.
Time Frame: From first dose of LCIG in this study up to 30 days after the date of last PEG-J exposure; median duration of treatment was 1178 days.
Population: All participants who received LCIG in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Participants
  Any device complication | 244
  Device complication leading to tube replacement | 183
  Device complication with associated adverse event | 177
  Device complication with associated adverse event leading to tube replacement | 43

3. Secondary Outcome: Number of Participants With Sleep Attacks
Description: Participants were asked whether they experienced any events in which they fell asleep suddenly or unexpectedly, including while engaged in some activity (e.g., eating/drinking, speaking, or driving) or at rest, with or without any previous warning of sleepiness. If yes, participants were asked if they suffered any "bad" outcome or problem from the falling asleep event.
Time Frame: Baseline (final assessment period of the previous open-label LCIG study) and every 6 months until final visit; median duration of treatment was 1178 days.
Population: All participants who received LCIG in this extension study with available sleep attack data. The number of participants who experienced a sleep attack with a bad outcome or problem is based on the number of participants who reported sleep attacks.
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Participants
  Baseline: One or more sleep attacks | 6
  Baseline: One or more sleep attacks with a bad outcome: number analyzed (Participants) | 6
  Baseline: One or more sleep attacks with a bad outcome | 0
  Post-baseline: One or more sleep attacks: number analyzed (Participants) | 255
  Post-baseline: One or more sleep attacks | 27
  Post-baseline: One or more sleep attacks with a bad outcome: number analyzed (Participants) | 27
  Post-baseline: One or more sleep attacks with a bad outcome | 3

4. Secondary Outcome: Number of Participants With Intense Impulsive Behavior
Description: To monitor for the development of intense impulsive behavior the Minnesota Impulsive Disorder Interview (MIDI) was administered. The MIDI is a semi-structured clinical interview assessing pathological gambling, trichotillomania, kleptomania, pyromania, intermittent explosive disorder, compulsive buying, and compulsive sexual behavior.
Time Frame: Baseline (final assessment of the previous open-label LCIG study) and every 6 months until final visit; median duration of treatment was 1178 days.
Population: All participants who received LCIG in this extension study with available MIDI data.
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Participants
  Baseline: Pathological Gambling | 1
  Baseline: Trichotillomania | 0
  Baseline: Kleptomania | 0
  Baseline: Pyromania | 0
  Baseline: Intermittent Explosive Disorder | 0
  Baseline: Compulsive Buying | 1
  Baseline: Compulsive Sexual Behavior | 1
  Post-baseline: Pathological Gambling: number analyzed (Participants) | 256
  Post-baseline: Pathological Gambling | 1
  Post-baseline: Trichotillomania: number analyzed (Participants) | 256
  Post-baseline: Trichotillomania | 0
  Post-baseline: Kleptomania: number analyzed (Participants) | 256
  Post-baseline: Kleptomania | 0
  Post-baseline: Pyromania: number analyzed (Participants) | 256
  Post-baseline: Pyromania | 0
  Post-baseline: Intermittent Explosive Disorder: number analyzed (Participants) | 256
  Post-baseline: Intermittent Explosive Disorder | 0
  Post-baseline: Compulsive Buying: number analyzed (Participants) | 256
  Post-baseline: Compulsive Buying | 2
  Post-baseline: Compulsive Sexual Behavior: number analyzed (Participants) | 256
  Post-baseline: Compulsive Sexual Behavior | 14

5. Secondary Outcome: Number of Participants Who Developed Melanoma
Description: A comprehensive assessment for the presence of melanoma was performed at least once a year by a dermatologist.
Time Frame: Once per year during the study; median duration of treatment was 1178 days.
Population: All participants who received LCIG in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Participants | 2

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (TE AESI)
Description: Adverse events of special interest (AESIs) were identified using standardized Medical Dictionary for Regulatory Activities (MedDRA) queries (SMQ) or company MedDRA queries (CMQs). The AESI in the following categories were identified on the basis of review of the clinical program and postmarketing observations where the treatment system is commercially available.
  * Procedure and device associated events
  * Polyneuropathy, included preferred terms in either the peripheral neuropathy or GuillainBarre syndrome standardized MedDRA query (narrow search), such as polyneuropathy, decreased vibratory sense, peripheral neuropathy, peripheral sensory neuropathy, neuralgia, demyelinating polyneuropathy, and sensory disturbance
  * Weight loss
  * Cardiovascular fatalities
  * Respiratory tract aspiration including aspiration pneumonia/pneumonitis.
Time Frame: as for outcome 1
Population: ll participants who received LCIG in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 262
Participants
  TE AESI related to procedure and device | 162
  TE AESI related to polyneuropathy | 24
  TE AESI related to weight loss | 53
  TE AESI related to cardiovascular fatalities | 7
  TE AESI related to aspiration | 71

7. Secondary Outcome: Number of Participants With Any Suicidal Ideation or Behavior
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) was implemented with Protocol Amendment 3 (20 March 2012) in order to assess suicidal behavior and ideation.
  Suicidal ideation includes the wish to be dead, nonspecific active suicidal thoughts, active ideation without intent to act, active ideation with some intent to act, and active ideation with specific plan or intent. Suicidal behavior includes actual attempts, interrupted attempts, aborted attempts, completed suicide, and preparatory acts or behaviors.
  The number of participants with affirmative responses on the C-SSRS at any time during the treatment period is reported.
Time Frame: Every 6 months (beginning with implementation of Protocol Amendment 3) until final visit; median duration of treatment was 1178 days.
Population: All participants who received LCIG in this extension study with available C-SSRS data.
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 210
Participants
  Any suicidal ideation or behavior | 32
  Any suicidal ideation | 30
  Any suicidal behavior | 6
  Non-suicidal self-injurious behavior | 1

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Values
Description: A vital sign value was considered potentially clinically significant if it satisfied the pre-specified criteria presented in the table and was also more extreme than the participant's corresponding Baseline value.
Time Frame: Baseline and every 6 months until final visit; median duration of treatment was 1178 days.
Population: All participants who received LCIG in this extension study with at least one post-baseline measurement for each parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 255
Participants
  Supine Systolic Blood Pressure ≥180 mmHg and > 40 mmHg increase from Baseline | 6
  Supine Systolic Blood Pressure ≤ 90 mmHg and > 30 mmHg decrease from Baseline | 13
  Standing Systolic Blood Pressure ≥ 180 mmHg and > 40 mmHg increase from Baseline: number analyzed (Participants) | 254
  Standing Systolic Blood Pressure ≥ 180 mmHg and > 40 mmHg increase from Baseline | 1
  Standing Systolic Blood Pressure ≤ 90 mmHg and > 30 mmHg decrease from Baseline: number analyzed (Participants) | 254
  Standing Systolic Blood Pressure ≤ 90 mmHg and > 30 mmHg decrease from Baseline | 26
  Orthostatic Change in Systolic Blood Pressure Decrease of ≥ 30 mmHg: number analyzed (Participants) | 253
  Orthostatic Change in Systolic Blood Pressure Decrease of ≥ 30 mmHg | 73
  Supine Diastolic Blood Pressure ≥ 105 mmHg and > 30 mmHg increase from Baseline | 2
  Supine Diastolic Blood Pressure ≤ 50 mmHg and > 30 mmHg decrease from Baseline | 6
  Standing Diastolic Blood Pressure ≥ 105 mmHg and > 30 mmHg increase from Baseline: number analyzed (Participants) | 254
  Standing Diastolic Blood Pressure ≥ 105 mmHg and > 30 mmHg increase from Baseline | 7
  Standing Diastolic Blood Pressure ≤ 50 mmHg and > 30 mmHg decrease from Baseline: number analyzed (Participants) | 254
  Standing Diastolic Blood Pressure ≤ 50 mmHg and > 30 mmHg decrease from Baseline | 14
  Orthostatic Change in Diastolic Blood Pressure Decrease of ≥ 20 mmHg: number analyzed (Participants) | 253
  Orthostatic Change in Diastolic Blood Pressure Decrease of ≥ 20 mmHg | 45
  Supine Pulse ≥ 120 bpm and > 30 bpm increase from Baseline | 0
  Supine pulse ≤ 50 bpm and > 30 bpm decrease from Baseline | 3
  Standing pulse ≥ 120 bpm and > 30 bpm increase from Baseline: number analyzed (Participants) | 254
  Standing pulse ≥ 120 bpm and > 30 bpm increase from Baseline | 5
  Standing pulse ≤ 50 bpm and > 30 bpm decrease from Baseline: number analyzed (Participants) | 254
  Standing pulse ≤ 50 bpm and > 30 bpm decrease from Baseline | 4
  Temperature ≥ 38.3℃ and ≥ 1.1℃ increase from Baseline: number analyzed (Participants) | 254
  Temperature ≥ 38.3℃ and ≥ 1.1℃ increase from Baseline | 0
  Weight ≥ 7% increase from Baseline: number analyzed (Participants) | 254
  Weight ≥ 7% increase from Baseline | 36
  Weight ≥ 7% decrease from Baseline: number analyzed (Participants) | 254
  Weight ≥ 7% decrease from Baseline | 140

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hematology Laboratory Values
Description: A laboratory value was considered potentially clinically significant if it satisfied the pre-specified criteria presented in the table and was also more extreme than the participant's corresponding Baseline value.
Time Frame: Baseline and every 6 months until final visit; median duration of treatment was 1178 days.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 196
Participants
  Red blood cells (RBC) < 2.0 × 10^12 cells/L (Female); < 2.5 × 10^12 cells/L (Male) | 0
  Haemoglobin < 90 g/L (Female); < 100 g/L (Male) | 9
  Haematocrit < 30% (Female); < 34% (Male): number analyzed (Participants) | 195
  Haematocrit < 30% (Female); < 34% (Male) | 16
  White blood cells (WBC) < 2.8 × 10^9 cells/L | 3
  WBC > 16.0 × 10^9 cells/L | 2
  Absolute neutrophil count < 1.2 × 10^9 cells/L: number analyzed (Participants) | 195
  Absolute neutrophil count < 1.2 × 10^9 cells/L | 2
  Lymphocytes > 80%: number analyzed (Participants) | 195
  Lymphocytes > 80% | 0
  Absolute lymphocyte count < 0.75 × 10^9 cells/L: number analyzed (Participants) | 195
  Absolute lymphocyte count < 0.75 × 10^9 cells/L | 14
  Eosinophils > 10%: number analyzed (Participants) | 195
  Eosinophils > 10% | 4
  Monocytes > 30%: number analyzed (Participants) | 195
  Monocytes > 30% | 1
  Platelet count < 95 × 10^9 cells/L: number analyzed (Participants) | 194
  Platelet count < 95 × 10^9 cells/L | 2
  Platelet count > 700 × 10^9 cells/L: number analyzed (Participants) | 194
  Platelet count > 700 × 10^9 cells/L | 0
  Mean corpuscular volume (MCV) < 60 fL: number analyzed (Participants) | 195
  Mean corpuscular volume (MCV) < 60 fL | 0
  MCV > 120 fL: number analyzed (Participants) | 195
  MCV > 120 fL | 0

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Chemistry Laboratory Values
Description: A laboratory value was considered potentially clinically significant if it satisfied the pre-specified criteria presented in the table and was also more extreme than the participant's corresponding baseline value.
  ULN = upper limit of normal
Time Frame: Baseline and every 6 months until final visit; median duration of treatment was 1178 days.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 198
Participants
  Creatinine > 177 µmol/L | 0
  Calcium < 1.75 mmol/L | 1
  Calcium > 3.0 mmol/L | 0
  Total bilirubin > 2 x ULN | 0
  Aspartate aminotransferase (AST) > 3 x ULN | 0
  Alanine aminotransferase (ALT) > 3 x ULN | 0
  Gamma glutamyl-transferase (GGT) > 3 x ULN | 5
  Lactate dehydrogenase (LDH) > 3 x ULN: number analyzed (Participants) | 197
  Lactate dehydrogenase (LDH) > 3 x ULN | 0
  Alkaline phosphatase (ALP) > 400 U/L | 0
  Creatine phosphokinase (CPK) > 3 x ULN | 6
  Non-fasting glucose < 2.78 mmol/L | 4
  Non-fasting glucose > 16.0 mmol/L | 1
  Uric acid > 500 µmol/L (Female); > 590 µmol/L (Male) | 0
  Blood urea nitrogen (BUN) > 10.8 mmol/L: number analyzed (Participants) | 95
  Blood urea nitrogen (BUN) > 10.8 mmol/L | 11
  Cholesterol > 12.9 mmol/L | 0

11. Secondary Outcome: Number of Participants With Vitamin Levels Outside of the Normal Range
Description: Special tests for vitamin deficiencies (folic acid, vitamin B6, vitamin B12, methylmalonic acid [MMA], and homocysteine) were implemented with Protocol Amendment 2 (27 July 2011). The number of participants with vitamin levels outside of the normal range at any time post-baseline is reported for each vitamin tested.
Time Frame: Every 6 months (beginning with implementation of Protocol Amendment 2) until final visit; median duration of treatment was 1178 days.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 214
Participants
  Vitamin B12 < 148 pmol/L: number analyzed (Participants) | 212
  Vitamin B12 < 148 pmol/L | 22
  Vitamin B12 > 775 pmol/L: number analyzed (Participants) | 212
  Vitamin B12 > 775 pmol/L | 46
  Methylmalonic acid > 0.4 µmol/L | 65
  Homocysteine < 3.7 µmol/L | 1
  Homocysteine > 13.9 µmol/L | 198
  Vitamin B6 < 20 nmol/L: number analyzed (Participants) | 211
  Vitamin B6 < 20 nmol/L | 155
  Vitamin B6 > 125 nmol/L: number analyzed (Participants) | 211
  Vitamin B6 > 125 nmol/L | 108
  Folic acid < 4.5 nmol/L: number analyzed (Participants) | 213
  Folic acid < 4.5 nmol/L | 6

12. Secondary Outcome: Number of Participants Receiving Concomitant Anti-Parkinson's Disease Medications by Treatment Year
Description: Participants could use oral levodopa-carbidopa for scheduled or supplemental bedtime/overnight doses after the pump was disconnected for the night, or as rescue medication in case of acute deterioration caused by failure of the LCIG system such as tubes and/or the pump or the onset of an acute illness.
  The initiation of additional concomitant PD medication was allowed at the discretion of the Investigator if medically indicated.
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10, > Year 10 (maximum time on treatment was approximately 11.5 years).
Population: Participants who received LCIG during each year in this extension study
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Participants who received LCIG during Year 1 of the extension study.
- Year 2: Participants who received LCIG during Year 2 of the extension study.
- Year 3: Participants who received LCIG during Year 3 of the extension study.
- Year 4: Participants who received LCIG during Year 4 of the extension study.
- Year 5: Participants who received LCIG during Year 5 of the extension study.
- Year 6: Participants who received LCIG during Year 6 of the extension study.
- Year 7: Participants who received LCIG during Year 7 of the extension study.
- Year 8: Participants who received LCIG during Year 8 of the extension study.
- Year 9: Participants who received LCIG during Year 9 of the extension study.
- Year 10: Participants who received LCIG during Year 10 of the extension study.
- > Year 10: Participants who received LCIG after Year 10 of the extension study.
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5 | Year 6 | Year 7 | Year 8 | Year 9 | Year 10 | > Year 10
Number analyzed (Participants) | 262 | 230 | 196 | 146 | 96 | 59 | 44 | 38 | 27 | 22 | 9
Participants
  No concomitant PD medications (LCIG only) | 126 | 107 | 96 | 74 | 52 | 38 | 33 | 28 | 21 | 17 | 8
  Concomitant oral levodopa/carbidopa | 100 | 91 | 74 | 55 | 37 | 16 | 9 | 8 | 5 | 4 | 1
  Other concomitant PD medications | 36 | 32 | 26 | 17 | 7 | 5 | 2 | 2 | 1 | 1 | 0

13. Secondary Outcome: Change in Average Daily "Off" Time Based on the Parkinson's Disease Symptom Diary at End of Treatment
Description: The PD symptom diary asks participants (or their caregivers) to indicate their status upon waking and every 30 minutes during their normal waking time according to the following categories: asleep, "off", "on" without dyskinesia, "on" with non-troublesome dyskinesia, or "on" with troublesome dyskinesia.
  "Off" time was defined as time when medication had worn off and was no longer providing benefit with regard to mobility, slowness, and stiffness.
  PD diary times were normalized to a 16-hour waking day and averaged for the 3 days prior to each study visit.
  A negative change for "off" time indicates improvement. The PD diary assessment was implemented with Protocol amendment 4 (December 2013) for participants at United States (US) sites only.
Time Frame: Prior to initial LCIG infusion (in the previous study, before the first LCIG infusion), Baseline (final assessment of the previous open-label LCIG study), and end of treatment; median duration of treatment was 1178 days.
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
hours
  Change from initial LCIG infusion | -3.97 (2.86)
  Change from Baseline | -0.19 (2.19)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel; Change from initial LCIG infusion to end of study in "off" time was assessed for significance using a 1-sample paired t test; Test type: Other; p < 0.001, One-sample t-test
Statistical Analysis 2: Comparison: Levodopa-Carbidopa Intestinal Gel; Change from Baseline to end of study in "off" time was assessed for significance using a 1-sample paired t-test; Test type: Other; p = 0.433, One-sample t-test

14. Secondary Outcome: Change in Average Daily "On" Time Without Troublesome Dyskinesia Based on the Parkinson's Disease Symptom Diary at End of Treatment
Description: The PD diary asks participants (or their caregivers) to indicate their status upon waking and every 30 minutes during their normal waking time according to the following categories: asleep, "off", "on" without dyskinesia, "on" with non-troublesome dyskinesia, or "on" with troublesome dyskinesia.
  "On" time is when medication is providing benefit with regard to mobility, slowness and stiffness. Dyskinesia is involuntary twisting, turning movements which are an effect of medication and occur during "on" time. Non-troublesome dyskinesia does not interfere with function or cause meaningful discomfort.
  "On" time without troublesome dyskinesia is the sum of "on" time without dyskinesia and "on" time with non-troublesome dyskinesia. PD diary times were normalized to a 16-hour waking day and averaged for the 3 days prior to each study visit. A positive change indicates improvement.
  The PD diary was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
hours
  Change from initial LCIG infusion | 3.86 (3.31)
  Change from Baseline | -0.51 (3.19)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel; Change from initial LCIG infusion to end of study in "on" time without troublesome dyskinesia was assessed for significance using a 1-sample paired t-test; Test type: Other; p < 0.001, One-sample t-test
Statistical Analysis 2: Comparison: Levodopa-Carbidopa Intestinal Gel; Change from Baseline to end of study in "on" time without troublesome dyskinesia was assessed for significance using a 1-sample paired t test; Test type: Other; p = 0.150, One-sample t-test

15. Secondary Outcome: Change in Average Daily "On" Time With Troublesome Dyskinesia Based on the Parkinson's Disease Symptom Diary at End of Treatment
Description: The PD diary asks participants (or their caregivers) to indicate their status upon waking and every 30 minutes during their normal waking time according to the following categories: asleep, "off", "on" without dyskinesia, "on" with non-troublesome dyskinesia, or "on" with troublesome dyskinesia.
  "On" time is when medication is providing benefit with regard to mobility, slowness and stiffness. Dyskinesia is involuntary twisting, turning movements which are an effect of medication and occur during "on" time. Troublesome dyskinesia interferes with function or causes meaningful discomfort.
  PD diary times were normalized to a 16-hour waking day and averaged for the 3 days prior to each study visit. A positive change indicates improvement.
  The PD diary was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
hours
  Change from initial LCIG infusion | 0.12 (3.03)
  Change from Baseline | 0.70 (2.66)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel; Change from initial LCIG infusion to end of study in "on" time with troublesome dyskinesia was assessed for significance using a 1-sample paired t test; Test type: Other; p = 0.725, One-sample t-test
Statistical Analysis 2: Comparison: Levodopa-Carbidopa Intestinal Gel; Change from Baseline to end of study in "on" time with troublesome dyskinesia was assessed for significance using a 1-sample paired t test; Test type: Other; p = 0.019, One-sample t-test

16. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score at End of Treatment
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of PD. It is made up of the following sections:
  I) Mentation, Behavior, and Mood;
  II) Activities of Daily Living;
  III) Motor Examinations;
  IV) Complications of Therapy sections (including dyskinesias).
  The Part I Score is the sum of the answers to the 4 questions that comprise Part I, each of which are measured on a 5-point scale (0-4). The Part I score ranges from 0-16 and higher scores are associated with more disability. A negative change from Baseline indicates improvement.
  The UPDRS was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
score on a scale
  Change from initial LCIG infusion: number analyzed (Participants) | 79
  Change from initial LCIG infusion | 1.51 (2.83)
  Change from Baseline | 1.46 (2.29)

17. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score at End of Treatment
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of PD. It is made up of the following sections:
  I) Mentation, Behavior, and Mood;
  II) Activities of Daily Living;
  III) Motor Examinations;
  IV) Complications of Therapy sections (including dyskinesias).
  The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability. A negative change from Baseline indicates improvement.
  The UPDRS was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
score on a scale
  Change from initial LCIG infusion: number analyzed (Participants) | 79
  Change from initial LCIG infusion | 3.04 (7.76)
  Change from Baseline | 6.11 (5.48)

18. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score at End of Treatment
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of PD. It is made up of the following sections:
  I) Mentation, Behavior, and Mood;
  II) Activities of Daily Living;
  III) Motor Examinations;
  IV) Complications of Therapy sections (including dyskinesias).
  UPDRS Part III consists of 14 questions. Questions 20 - 26 are multi-part questions in that they are evaluated separately for multiple body parts. Counting each of these assessments leads to a total of 27 answers for Part III. The UPDRS Part III score is the sum of the 27 answers provided to the 14 Part III questions, each of which are measured on a 5-Point scale (0-4). The Part III score ranges from 0-108 and higher scores are associated with more disability. A negative change from Baseline indicates improvement.
  The UPDRS was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
score on a scale
  Change from initial LCIG infusion: number analyzed (Participants) | 79
  Change from initial LCIG infusion | 4.51 (14.71)
  Change from Baseline | 9.18 (10.63)

19. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score at End of Treatment
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of PD. It is made up of the following sections:
  I) Mentation, Behavior, and Mood;
  II) Activities of Daily Living;
  III) Motor Examinations;
  IV) Complications of Therapy sections (including dyskinesias).
  The UPDRS total score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I - III of the scale. The total score ranges from 0 - 176 with 176 representing the worst (total) disability, and 0 no disability. A negative change from Baseline indicates improvement.
  The UPDRS was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
score on a scale
  Change from initial LCIG infusion: number analyzed (Participants) | 79
  Change from initial LCIG infusion | 9.12 (20.91)
  Change from Baseline | 16.82 (15.01)

20. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Score at End of Treatment
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of PD. It is made up of the following sections:
  I) Mentation, Behavior, and Mood;
  II) Activities of Daily Living;
  III) Motor Examinations;
  IV) Complications of Therapy sections (including Dyskinesias).
  The UPDRS Part IV Score is the sum of all answers to the 11 questions that comprise Part IV, 4 of which are measured on a 5-point scale (0 - 4) and 7 which are measured on a 2-point scale (0 - 1). The Part IV score ranges from 0 - 23 with higher scores associated with more disability. A negative change from Baseline indicates improvement.
  The UPDRS was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
score on a scale
  Change from initial LCIG infusion: number analyzed (Participants) | 79
  Change from initial LCIG infusion | -2.27 (3.70)
  Change from Baseline | 0.77 (2.86)

21. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Dyskinesia Score at End of Treatment
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of PD. It is made up of the following sections:
  I) Mentation, Behavior, and Mood; II) Activities of Daily Living; III) Motor Examinations; IV) Complications of Therapy sections (including Dyskinesias); and
  The UPDRS Part IV dyskinesia Score is the sum of Questions 32 (What proportion of the waking day are dyskinesias present?), 33 (How disabling are the dyskinesias? ), and 34 (How painful are the dyskinesias?) on UPDRS Part IV, each of which are measured on a 5-point scale (0-4). The Part IV dyskinesia score ranges from 0 - 12 and higher scores are associated with more disability. A negative change from Baseline indicates improvement.
  The UPDRS was implemented with Protocol amendment 4 (December 2013) for participants at US sites only.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 82
score on a scale
  Change from initial LCIG infusion: number analyzed (Participants) | 79
  Change from initial LCIG infusion | -0.19 (2.55)
  Change from Baseline | 0.55 (1.86)

22. Secondary Outcome: Change in Parkinson's Disease Questionnaire (PDQ-39) Scores at End of Treatment
Description: The PDQ-39 is a self-administered questionnaire that comprises 39 items addressing the following eight domains of health that patients consider to be adversely affected by the disease:
  * Mobility (e.g., fear of falling when walking) - 10 questions
  * Activities of daily living (e.g., difficulty cutting food) - 6 questions
  * Emotional well-being (e.g., feelings of isolation) - 6 questions
  * Stigma (e.g., social embarrassment) - 4 questions
  * Social support - 3 questions
  * Cognition - 4 questions
  * Communication - 3 questions
  * Bodily discomfort - 3 questions
  Each question is answered on a 5-point scale from 0 (Never) to 4 (Always / Cannot Do At All). Scores are calculated by summing the answers to the questions in the domain and converting to a scale from 0 to 100. Higher scores are associated with the more severe symptoms of the disease such as tremor and stiffness. The PDQ-39 summary index (range 0-100) includes responses to all 39 items. A negative change indicates improvement.
Time Frame: as for outcome 13
Population: Participants who were enrolled in the United States and had at least 1 efficacy assessment in the current study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 102
score on a scale
  Summary Index: Change from initial LCIG infusion | -1.46 (16.98)
  Summary Index: Change from Baseline | 6.83 (13.14)
  Mobility Domain: Change from initial LCIG infusion | -2.08 (27.98)
  Mobility Domain: Change from Baseline | 12.01 (21.81)
  Activities of Daily Living Domain: Change from initial LCIG infusion | -1.55 (28.40)
  Activities of Daily Living Domain: Change from Baseline | 9.35 (20.40)
  Emotional Well-Being Domain: Change from initial LCIG infusion: number analyzed (Participants) | 101
  Emotional Well-Being Domain: Change from initial LCIG infusion | -0.58 (19.31)
  Emotional Well-Being Domain: Change from Baseline | 2.53 (16.95)
  Stigma Domain: Change from initial LCIG infusion | -9.50 (22.49)
  Stigma Domain: Change from Baseline | -0.18 (19.52)
  Social Support Domain: Change from initial LCIG infusion: number analyzed (Participants) | 101
  Social Support Domain: Change from initial LCIG infusion | 3.59 (19.54)
  Social Support Domain: Change from Baseline | 2.25 (17.88)
  Cognition Domain: Change from initial LCIG infusion | 1.78 (19.52)
  Cognition Domain: Change from Baseline | 6.56 (19.63)
  Communication Domain: Change from initial LCIG infusion | 3.19 (23.01)
  Communication Domain: Change from Baseline | 8.17 (19.27)
  Bodily Discomfort Domain: Change from initial LCIG infusion | -4.74 (24.61)
  Bodily Discomfort Domain: Change from Baseline | 5.64 (19.70)

ADVERSE EVENTS:
Time Frame: From first dose of LCIG in this study up to 30 days after the date of last PEG-J exposure; median duration of treatment was 1178 days, and maximum was 4217 days (11.5 years).
Arm/Group | Levodopa-Carbidopa Intestinal Gel
All-Cause Mortality (participants affected / at risk) | 59/262
Serious Adverse Events (participants affected / at risk) | 159/262
Other Adverse Events (participants affected / at risk) | 223/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (N=262)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 3 (3)
CARDIAC FAILURE (Cardiac disorders) | 2 (2)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 3 (3)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (2)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1)
EXTRASYSTOLES (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4)
SICK SINUS SYNDROME (Cardiac disorders) | 2 (2)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
VENOUS STASIS RETINOPATHY (Eye disorders) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (5)
BEZOAR (Gastrointestinal disorders) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 3 (5)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 4 (4)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2)
GIANT CELL EPULIS (Gastrointestinal disorders) | 1 (1)
ILEUS PARALYTIC (Gastrointestinal disorders) | 2 (2)
INGUINAL HERNIA (Gastrointestinal disorders) | 3 (3)
INTESTINAL DILATATION (Gastrointestinal disorders) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3)
INTUSSUSCEPTION (Gastrointestinal disorders) | 2 (2)
JEJUNAL ULCER (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (2)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 3 (3)
PERITONITIS (Gastrointestinal disorders) | 1 (1)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 2 (2)
RECTAL PROLAPSE (Gastrointestinal disorders) | 2 (2)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOLVULUS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2)
ASTHENIA (General disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
COMPLICATION OF DEVICE INSERTION (General disorders) | 14 (24)
DEATH (General disorders) | 13 (13)
DEVICE BREAKAGE (General disorders) | 1 (1)
DEVICE DISLOCATION (General disorders) | 6 (8)
DEVICE MATERIAL ISSUE (General disorders) | 1 (1)
DEVICE OCCLUSION (General disorders) | 1 (3)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2)
MALAISE (General disorders) | 1 (1)
MEDICAL DEVICE SITE REACTION (General disorders) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 2 (2)
NECROSIS (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
PYREXIA (General disorders) | 2 (2)
SUDDEN DEATH (General disorders) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (3)
CORONA VIRUS INFECTION (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
GANGRENE (Infections and infestations) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 20 (23)
POST PROCEDURAL SEPSIS (Infections and infestations) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 9 (11)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1)
PYOTHORAX (Infections and infestations) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6)
WOUND INFECTION (Infections and infestations) | 1 (1)
WOUND INFECTION PSEUDOMONAS (Infections and infestations) | 1 (1)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (2)
FALL (Injury, poisoning and procedural complications) | 13 (15)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 4 (5)
HEAD INJURY (Injury, poisoning and procedural complications) | 2 (2)
HEAT STROKE (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 5 (5)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PERIPROSTHETIC OSTEOLYSIS (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 1 (1)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)
BLOOD MAGNESIUM DECREASED (Investigations) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1)
HAEMATOCRIT DECREASED (Investigations) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1)
HEART RATE DECREASED (Investigations) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
URINE OUTPUT DECREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 8 (10)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1)
VITAMIN B6 DEFICIENCY (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CAMPTOCORMIA (Musculoskeletal and connective tissue disorders) | 1 (1)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (5)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PERIPHERAL T-CELL LYMPHOMA UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BALANCE DISORDER (Nervous system disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 2 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (3)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 2 (2)
DEMENTIA (Nervous system disorders) | 2 (2)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 2 (2)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 3 (5)
MENTAL IMPAIRMENT (Nervous system disorders) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
MONOPLEGIA (Nervous system disorders) | 1 (1)
MYOCLONUS (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
ON AND OFF PHENOMENON (Nervous system disorders) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 8 (8)
PARKINSONIAN CRISIS (Nervous system disorders) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 2 (2)
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 (1)
SCIATICA (Nervous system disorders) | 1 (1)
SEDATION (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 4 (5)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 2 (2)
AFFECTIVE DISORDER (Psychiatric disorders) | 1 (1)
AGGRESSION (Psychiatric disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (3)
DELIRIUM (Psychiatric disorders) | 2 (2)
DOPAMINE DYSREGULATION SYNDROME (Psychiatric disorders) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 2 (2)
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 3 (3)
PARANOIA (Psychiatric disorders) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1)
SLEEP ATTACKS (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 2 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2)
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (2)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 (2)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 3 (3)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1)
PELVIC HAEMATOMA (Reproductive system and breast disorders) | 1 (1)
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 9 (12)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 5 (5)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 3 (3)
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 2 (2)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1)
SUBGALEAL HAEMATOMA (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (N=262)
ANAEMIA (Blood and lymphatic system disorders) | 18 (21)
CATARACT (Eye disorders) | 13 (17)
ABDOMINAL PAIN (Gastrointestinal disorders) | 22 (27)
CONSTIPATION (Gastrointestinal disorders) | 30 (39)
DIARRHOEA (Gastrointestinal disorders) | 24 (29)
NAUSEA (Gastrointestinal disorders) | 32 (40)
COMPLICATION OF DEVICE INSERTION (General disorders) | 19 (25)
FATIGUE (General disorders) | 15 (17)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 55 (95)
URINARY TRACT INFECTION (Infections and infestations) | 45 (86)
FALL (Injury, poisoning and procedural complications) | 47 (70)
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 38 (46)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 24 (31)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 28 (39)
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 33 (47)
BLOOD HOMOCYSTEINE INCREASED (Investigations) | 59 (64)
VITAMIN B6 DECREASED (Investigations) | 71 (98)
VITAMIN B6 INCREASED (Investigations) | 21 (25)
WEIGHT DECREASED (Investigations) | 32 (36)
VITAMIN B6 DEFICIENCY (Metabolism and nutrition disorders) | 20 (22)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 22 (31)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21 (24)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 15 (20)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (22)
BALANCE DISORDER (Nervous system disorders) | 14 (17)
COGNITIVE DISORDER (Nervous system disorders) | 18 (18)
DYSKINESIA (Nervous system disorders) | 28 (34)
PARKINSON'S DISEASE (Nervous system disorders) | 28 (38)
ANXIETY (Psychiatric disorders) | 24 (27)
DEPRESSION (Psychiatric disorders) | 32 (35)
HALLUCINATION (Psychiatric disorders) | 17 (20)
INSOMNIA (Psychiatric disorders) | 31 (35)
SLEEP ATTACKS (Psychiatric disorders) | 16 (19)
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 41 (67)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2013-12-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT00660673/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT00660673/SAP_001.pdf